CLINICAL TRIAL: NCT00747461
Title: Assessment of the Safety, Side Effects and Efficacy of Interventional Cryotherapy for the Eradication of Benign Airway Disease("ICE THE BAD")
Brief Title: Interventional Cryotherapy for the Eradication of Benign Airway Disease ("ICE the BAD")
Acronym: ICEtheBAD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00026
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Results first posted 2015-06-26 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Lung Diseases, Obstructive; Sarcoidosis; Wegener's Granulomatosis; Rhinoscleroma; Recurrent Respiratory Papillomatosis
Keywords: Benign Airway Disease; Airway Injury; Sarcoidosis; Wegener's Granulomatosis; Rhinoscleroma; Recurrent Respiratory Papillomatosis(RRP)
MeSH Terms: conditions — Lung Diseases, Obstructive; Sarcoidosis; Granulomatosis with Polyangiitis; Rhinoscleroma; Recurrent respiratory papillomatosis | interventions — Cryotherapy; Cryosurgery; Cryoelectron Microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryospray Ablation (Experimental): Experimental CSA (Cryospray Ablation)
  Interventions: Device: CryoSpray Ablation

INTERVENTIONS:
Device: CryoSpray Ablation — Cryospray Ablation up to 4 -5 second cycles for up to 4 treatments in the first 30 days
  Other Names: CryoSpray Ablation(TM)System; Cryotherapy; Cryosurgery; Cryospray; Cryo

SUMMARY:
The purpose of this study is to evaluate the safety, effectiveness, and side effects of the CryoSpray AblationTM System (CryoSpray AblationTM, "CSA" or "cryospray therapy") to treat benign airway disease in the lung using liquid nitrogen sprayed through a catheter via flexible fiber optic bronchoscopy (FFB)

DETAILED DESCRIPTION:
The proposed study is a single center pilot study consisting of up to 10 subjects with benign airway disease. Treatment dosimetry will be up to 4, 5-second spray cycles. Subjects will have initial cryospray treatment at Day 0. Subjects will undergo repeat bronchoscopy in the first three to seven days after the initial treatment, to check for mucosal sloughing and to reassess luminal patency of the airway. Subjects may undergo up to one bronchoscopy per week with CSA therapy for a total of four (4) treatments in the first month. If they present with symptoms thereafter, then a repeat bronchoscopy will be performed; if luminal obstruction is noted, then the subject will begin the treatment protocol again. If disease exists bilaterally, only one side will be sprayed initially.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Deemed a candidate for cryotherapy based on physician physical or medical history review
* Deemed operable based on institutional criteria.

Exclusion Criteria:

* Pregnant or nursing
* Planning to sire a child while enrolled in the study
* Known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines.
* Refusal or inability to give consent.
* Concurrent chemotherapy.
* Prior radiation therapy which involved the any area between the vocal chords and the diaphragm
* Medical contraindication or potential problem that would preclude study participation
* Concurrent participation in other experimental studies Uncontrolled coagulopathy or bleeding diathesis

Serious medical illness, including:

* Uncontrolled congestive heart failure
* Uncontrolled angina
* Myocardial infarction
* Cerebrovascular accident within 6 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Machuzak, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Johnston MH, Eastone JA, Horwhat JD, Cartledge J, Mathews JS, Foggy JR. Cryoablation of Barrett's esophagus: a pilot study. Gastrointest Endosc. 2005 Dec;62(6):842-8. doi: 10.1016/j.gie.2005.05.008. PMID 16301023
- [Background] Johnston CM, Schoenfeld LP, Mysore JV, Dubois A. Endoscopic spray cryotherapy: a new technique for mucosal ablation in the esophagus. Gastrointest Endosc. 1999 Jul;50(1):86-92. doi: 10.1016/s0016-5107(99)70352-4. PMID 10385730
- [Background] Ell C, May A, Gossner L, Pech O, Gunter E, Mayer G, Henrich R, Vieth M, Muller H, Seitz G, Stolte M. Endoscopic mucosal resection of early cancer and high-grade dysplasia in Barrett's esophagus. Gastroenterology. 2000 Apr;118(4):670-7. doi: 10.1016/s0016-5085(00)70136-3. PMID 10734018
- [Background] Champion G, Richter JE, Vaezi MF, Singh S, Alexander R. Duodenogastroesophageal reflux: relationship to pH and importance in Barrett's esophagus. Gastroenterology. 1994 Sep;107(3):747-54. doi: 10.1016/0016-5085(94)90123-6. PMID 8076761
- [Background] Eisen GM, Sandler RS, Murray S, Gottfried M. The relationship between gastroesophageal reflux disease and its complications with Barrett's esophagus. Am J Gastroenterol. 1997 Jan;92(1):27-31. PMID 8995932
- [Background] Johnston MH. Cryotherapy and other newer techniques. Gastrointest Endosc Clin N Am. 2003 Jul;13(3):491-504. doi: 10.1016/s1052-5157(03)00044-8. PMID 14629105
- [Background] Cash BD, Johnston LR, Johnston MH. Cryospray ablation (CSA) in the palliative treatment of squamous cell carcinoma of the esophagus. World J Surg Oncol. 2007 Mar 16;5:34. doi: 10.1186/1477-7819-5-34. PMID 17367523
- [Background] Field JK, Youngson JH. The Liverpool Lung Project: a molecular epidemiological study of early lung cancer detection. Eur Respir J. 2002 Aug;20(2):464-79. doi: 10.1183/09031936.02.00290202. PMID 12212983
- [Background] Pinsonneault C, Fortier J, Donati F. Tracheal resection and reconstruction. Can J Anaesth. 1999 May;46(5 Pt 1):439-55. doi: 10.1007/BF03012943. PMID 10349923
- [Background] Dumot JA. Cryotherapy Ablation for Esophageal HGD or IMCA in High Risk, Non-Surgical Patients. DDW2007 Abstract submission. Cleveland Clinic Foundation (pending publication)
- [Background] Greenwald BD. CryoSpray Ablation of Early Esophageal Cancer. DDW 2007 Abstract submission. University of Maryland Medical Center. (pending publication)
- [Background] Johnston M, Horwhat J, Dubois A, Schoenfeld P. Endoscopic cryotherapy in the swine esophagus: A follow-up study (Abstract). Gastrointestinal Endoscopy 49:AB126, 1999.
- [Background] Johnston MH, Horwhat JD, Haluska, Moses FM. Depth of injury following endoscopic spray cryotherapy: EUS assisted evaluation of mucosal ablation and subsequent healing in the swine model (Abstract). Gastrointestinal Endoscopy 51: AB98, 3462, 2000.
- [Background] Johnston MH. Endoscopic cryotherapy: A new ice age in gastroenterology? Medscape Gastroenterology 2: 187, 2000.
- [Background] Eastone JA, Horwhat D, Haluska O, Mathews J, Johnston M. Cryoablation of swine esophageal mucosa: A direct comparison to argon plasma coagulation (APC) and multipolar electrocoagulation (MPEC) [Abstract] Gastrointestinal Endoscopy 53: A3448, 2001.
- [Background] Johnston MH, Eastone JA, Horwhat JD. Reversal of Barrett's esophagus with cryotherapy [Abstract]. American Journal of Gastroenterology 98(9 Suppl): A30, S11, 2003.
- [Background] Johnston MH, Cash BD, Horwhat JD, Johnston LR, Dykes CA, Mays HS. Cryoablation of Barrett's Esophagus (BE) [Abstract]. Gastroenterology 130 (4, Suppl.2): A640, 2006.
- [Background] Johnston MH, Cash BD, Dykes CA, Mays HS, Johnston LR. Cryoablation of dysplasia in Barrett's Esophagus (BE) and early stage esophageal cancer [Abstract]. Gastrointestinal Endoscopy 63 (5): April, 2006.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cryo Spray Ablation: subjects receiving up to 4 -5 second spray cycles
Period: Overall Study
Arm/Group | Cryo Spray Ablation
Started | 5
Completed | 0
Not Completed | 5
Not completed — study terminated by sponsor | 5

BASELINE CHARACTERISTICS:
Groups:
- Cryo Spray Ablation: subjects will receive up to 4 -5 second cycles of cryospray ablation
Arm/Group | Cryo Spray Ablation
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Luminal Patency Following Cryospray Treatment
Time Frame: 30 days
Population: study terminated by Sponsor-data not analyzed
Groups:
- Cryo Spray Ablation: Subject receiving cryo spray ablation
Arm/Group | Cryo Spray Ablation
Number analyzed (Participants) | 0

2. Secondary Outcome: Treatment Durability
Description: need for additional treatments within specified period
Time Frame: 12 months
Population: study terminated-no subjects analyzed.
Groups:
- Cryo Spray Ablation: subjects receiving cryo spray ablation
Arm/Group | Cryo Spray Ablation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- All Subjects Receiving CSA Cryospray: All subjects enrolled will received CSA cryospray.
  CryoSpray Ablation (tm): The CryoSpray Ablation(TM) System is a cryosurgical device utilizing a low-pressure liquid nitrogen spray tip CSATM Catheter. Medical grade liquid nitrogen is the cryogen used in the device. The device is used to destroy unwanted tissue by the application of extreme cold with the focused application to select tissue. The cryogen is stored in a liquid nitrogen holding tank integrated into the system.
Arm/Group | All Subjects Receiving CSA Cryospray
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No